CLINICAL TRIAL: NCT04906382
Title: Pilot Study of Tislelizumab (BGB-A317) in Recurrent Mismatch Repair Deficient Endometrial Cancer and the Effect on the Tumor Microenvironment
Brief Title: Tislelizumab for the Treatment of Recurrent Mismatch Repair Deficient Endometrial Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor reorganization
Sponsor: Floor Backes, MD (Other)
Responsible Party: Sponsor-Investigator, Floor Backes, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20173; NCI-2021-01367 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-03-22; First posted 2021-05-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Lynch Syndrome; Recurrent Endometrial Carcinoma; Recurrent Endometrial Clear Cell Adenocarcinoma; Recurrent Uterine Corpus Carcinosarcoma; Mismatch Repair Deficiency; Recurrent Endometrial Cancer; Metastatic Endometrial Cancer
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms; Turcot syndrome | interventions — Biopsy; Carboplatin; Paclitaxel; Taxes; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tislelizumab) (Experimental): Chemo naïve patients receive tislelizumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Beginning cycle 4, patients who are chemotherapy naive with progressive disease, stable disease, or partial response, also receive carboplatin IV and paclitaxel IV every 21 days per standard of care for 6-9 cycles at the discretion of the treating physician.
  Patients who have received prior chemotherapy will receive single agent tislelizumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Drug: Carboplatin; Drug: Paclitaxel; Biological: Tislelizumab

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Tislelizumab — Given IV
  Other Names: BGB-A317

SUMMARY:
This clinical trial evaluates the effect of tislelizumab in treating patients with mismatch repair deficient endometrial cancer that has come back (recurrent). Deoxyribonucleic acid (DNA) mismatch repair (MMR) is a system for recognizing and repairing DNA errors and damage. Mismatch repair deficient tumors (dMMR) may have difficulty repairing DNA mutations during replication that may affect tumor's response to therapy. Immunotherapy with monoclonal antibodies, such as tislelizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving tislelizumab may help treat patients with mismatch repair deficient endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of tislelizumab (BGB-A317) on the diversity and dynamics of the T cell receptor repertoire in responders versus non-responders.

SECONDARY OBJECTIVES:

I. To evaluate the effect of tislelizumab on tumor mutational profiles between responders and non-responders.

II. To evaluate the effect of tislelizumab +/- carboplatin/paclitaxel on PD-1/PD-L1 expression and other immune markers in tumor biopsies between responders and non-responders.

III. To evaluate the safety and tolerability of tislelizumab +/- carboplatin/paclitaxel in patients with MMR deficient recurrent endometrial cancer.

EXPLORATORY OBJECTIVES:

I. To explore the effect of adding carboplatin/paclitaxel to tislelizumab on tumor mutational profiles.

II. To explore the effect of adding carboplatin/paclitaxel to tislelizumab (BGB-A317) on the diversity and dynamics of the T cell receptor repertoire.

III. To explore the objective antitumor activity (complete and partial response) of tislelizumab as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria.

IV. To explore the objective antitumor activity (complete and partial response) of tislelizumab/carboplatin/paclitaxel after single agent tislelizumab as measured by RECIST v1.1 criteria V. To explore the progression free survival in patients with mismatch repair deficiency (dMMR) recurrent endometrial cancer treated with tislelizumab +/- carboplatin/paclitaxel.

OUTLINE:

Patients receive tislelizumab intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Beginning cycle 4, patients who are chemotherapy naive with progressive disease, stable disease, or partial response, also receive carboplatin IV and paclitaxel IV every 21 days per standard of care for 6-9 cycles at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 30, 60, and 90 days, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
* Age >= 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
* All patients with recurrent endometrial carcinoma, of any histology including clear cell, serous papillary carcinomas, and carcinosarcoma, whose disease is not amenable to definitive local therapy (including surgery and/or radiation therapy)
* Patients must have deficient mismatch repair as demonstrated by lack of expression of at least 1 mismatch repair protein by immunohistochemistry, or evidence of microsatellite instability (MSI) high, or evidence of Lynch syndrome
* The patient must have a lesion that is amenable to safe biopsy and the patient must agree to pre-and post-treatment biopsies
* Patients may have received radiation for the treatment of endometrial cancer
* Patient must have recovered from toxicity related to prior treatment to grade 2 or less
* At least two weeks should have elapsed since completion of prior chemotherapy or 5 half-lives (whichever is shorter), or 4 weeks from radiation involving the whole pelvis or over 50% of the spine
* At least 1 measurable lesion as defined per RECIST v1.1 that is amenable to biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (must not have required a blood transfusion or growth factor support =< 14 days before sample collection at screening) (during screening or =< 14 days prior to first dose of study drug)
* Platelets >= 75 x 10^9/L (must not have required a blood transfusion or growth factor support =< 14 days before sample collection at screening) (during screening or =< 14 days prior to first dose of study drug)
* Hemoglobin >= 9.0 g/dL (must not have required a blood transfusion or growth factor support =< 14 days before sample collection at screening) (during screening or =< 14 days prior to first dose of study drug)
* Serum creatinine =< 1.5 x ULN (upper limit of normal) or estimated glomerular filtration rate >= 30 mL/min/1.73 m^2 by Chronic Kidney Disease Epidemiology Collaboration equation (during screening or =< 14 days prior to first dose of study drug)
* Serum total bilirubin =< 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome) (during screening or =< 14 days prior to first dose of study drug)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (during screening or =< 14 days prior to first dose of study drug)
* Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and >= 120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test =< 7 days of first dose of study drug

Exclusion Criteria:

* Prior therapies targeting PD-1 or PD-L1
* Patients with symptomatic pleural effusion are excluded
* Active leptomeningeal disease or uncontrolled brain metastasis.

  * Following treatment, these patients may then be eligible, provided all other criteria, including those for patients with a history of brain metastases, are met
* Active autoimmune diseases or history of autoimmune diseases that may relapse.
* Any active malignancy =< 2 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
* Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication =< 14 days before first dose of study drug
* With uncontrolled diabetes or laboratory test abnormalities > grade 1 in potassium, sodium, or corrected calcium despite standard medical management or >= grade 3 hypoalbuminemia =< 14 days before first dose of study drug
* With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
* With severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy within 14 days prior to randomization or first dose of study drugs
* Human immunodeficiency virus (HIV) testing is not required by protocol unless clinically indicated. Known HIV positive patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; and cirrhosis. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Any major surgical procedure requiring general anesthesia =< 28 days before first dose of study drug
* Prior allogeneic stem cell transplantation or organ transplantation
* Any of the following cardiovascular risk factors:

  * Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, =< 28 days before first dose of study drug
  * Symptomatic pulmonary embolism =< 28 days before first dose of study drug
  * Any history of acute myocardial infarction =< 6 months before first dose of study drug
  * Any history of heart failure meeting New York Heart Association (NYHA) classification III or IV =< 6 months before first dose of study drug
  * Any event of ventricular arrhythmia >= grade 2 in severity =< 6 months before first dose of study drug
  * Any history of cerebrovascular accident =< 6 months before first dose of study drug
  * Uncontrolled hypertension: systolic pressure >= 160 mmHg or diastolic pressure >= 100 mmHg despite anti-hypertension medications =< 28 days before randomization or first dose of drug
  * Any episode of syncope or seizure =< 28 days before first dose of study drug
* A history of severe hypersensitivity reactions to tislelizumab
* Has received any chemotherapy, immunotherapy (e.g., interleukin, interferon, thymoxin) or any investigational therapies within 14 days or 5 half-lives (whichever is shorter) of the first study drug administration
* Has received any herbal medicine used to control cancer within 14 days of the first study drug administration
* Was administered a live vaccine =< 4 weeks before first dose of study drug

  * Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines, and are not allowed
* Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct
* Concurrent participation in another therapeutic clinical study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
T-cell receptor (TCR) profiles | Up to 24 months
  1) Measurements of TCRB clonal expansion in peripheral blood. Measurements of TCR in peripheral blood/-tissue
T-cell receptor (TCR) clonality | Up 24 month
  Measurements of TCRB clonal expansion in peripheral blood.
T-cell receptor (TCR) diversity | Up to 24 months
  Measurements of TCRB diversity in peripheral blood

SECONDARY OUTCOMES:
Tumor mutational profiles | Up to 3 years
  Evaluated using whole exome sequencing
PD-L1 expression and other immune markers in tissue | up to 24 weeks
  Evaluated using immunohistochemistry
Overall response rate (objective response rate complete response [CR] and partial response [PR]; clinical benefit rate CR + PR + stable) | Up to 3 years
  Evaluated by Response Evaluation Criteria in Solid Tumors version 1.1.
Progression-free survival | From date of enrollment to date of progressive disease, assessed up to 5 years
  Estimated using Kaplan-Meier method.
Overall survival | Up to 5 years
  Estimated using Kaplan-Meier method.
Incidence of adverse events | Up to 2 years
  Assessed using CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Floor Backes, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT04906382/ICF_000.pdf